CLINICAL TRIAL: NCT04128969
Title: Causal Mechanisms in Adolescent Arterial Stiffness
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Justin Zachariah, Principal Investigator. Assistant Professor in Pediatrics, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-45557; R01HL148217 (NIH)
Record Dates: First submitted 2019-10-11; First posted 2019-10-16 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Lipid Disorder; Dyslipidemias; Aortic Stiffness; Insulin Resistance Syndrome; Metabolic Syndrome; Pediatric Obesity
Keywords: dyslipidemia; arterial stiffness; pediatric obesity; metabolic syndrome; insulin resistance
MeSH Terms: conditions — Lipid Metabolism Disorders; Dyslipidemias; Metabolic Syndrome; Pediatric Obesity; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carnitine supplementation (CS+) (Experimental): Carnitine supplementation in liquid form, sugar free.
  Interventions: Dietary Supplement: CS+
- Placebo (CS-) (Placebo Comparator): Placebo comparator liquid similar in appearance and taste to CS+.
  Interventions: Dietary Supplement: CS-

INTERVENTIONS:
Dietary Supplement: CS+ — Oral carnitine supplementation
  Arms: Carnitine supplementation (CS+)
Dietary Supplement: CS- — Placebo
  Arms: Placebo (CS-)

SUMMARY:
Hardening of the blood vessels, called arterial stiffness, is a risk factor for future heart disease and its causes are unclear. The proposed study will 1) randomly assign adolescents at high risk of stiffening blood vessels to take a protein supplement called carnitine and study its effects on arterial stiffening and 2) study carnitine related genes for their effect on arterial stiffening. The study will definitively establish a role for carnitine action as a cause of stiffening blood vessels and signal a way to treat or prevent stiffening.

DETAILED DESCRIPTION:
Aortic stiffness measured in adolescence or adulthood determines current hypertension, predicts future incidence of hypertension, and future atherosclerotic cardiovascular disease (ASCVD) events. International hypertension guidelines list severe aortic stiffness as grounds to intensify anti-hypertensive pharmacotherapy. Mechanisms of arterial stiffness beyond aging and obesity warrant further elucidation. In our preliminary data from adolescents attending weight-loss summer camps arterial stiffness improvement was not associated with weight change but was with change in circulating carnitine. Carnitine influences fatty acid oxidation and carbohydrate metabolism. Carnitine could therefore link to arterial stiffness through insulin resistance which in turn affects cellular tone, vascular fibrosis, modification of lipids or glucose metabolism, and/or advanced glycation end products. This proposal leverages 2 instrumental variable study designs to infer a causal relation between carnitine and arterial stiffness. First, in 90 youth 11-21 years old at risk of arterial stiffening due to high serum triglycerides(TG), we will conduct a mechanistic, double blinded, randomized controlled trial for the effect of 6 months of oral carnitine supplementation (CS+, n=45) versus placebo (CS-, n=45) on aortic stiffness measured as carotid femoral pulse wave velocity (CFPWV); serum fatty acid oxidation biomarkers by metabolomics analysis; insulin resistance as homeostatic model assessment of insulin resistance (HOMA-IR); and TG. Aim 1 is to compare CS+ versus CS- on change in arterial stiffness and monitor adverse events. The hypothesis CS+ is associated with lower arterial stiffening, and CS+ effect is not modified by sex or race/ethnicity. Aim 2 is to compare the effect of CS+ versus CS- on fatty acid metabolism, insulin resistance, and lipids. The hypothesis is that CS+ alters long chain fatty acid beta oxidation, measured as lower long chain acylcarnitines, which in turn improves (HOMA-IR), and in turn decreases TG levels. This causal chain will be disentangled for direct versus indirect effects on CFPWV change. Second, naturally randomly assorted carnitine single nucleotide polymorphisms (SNPs) noted above will be used to characterize the relationship of carnitine to arterial stiffness and stratify the effectiveness of CS+.Aim 3a is to obtain the direct effect of carnitine on arterial stiffness using Mendelian randomization of SNPs associated with serum carnitine as instrumental variables with the hypothesis these variant SNPs are associated with lower arterial stiffness, supporting a causal inference. Aim 3b is to identify effect modification of CS+ vs CS- on arterial stiffness by examining if a carnitine genetic risk score will modify the effect of CS+ on change in arterial stiffness. This proposal with 2 instrumental variable projects would evaluate a causal role for carnitine in arterial stiffness at a point when the life course trajectory to hypertension can be modified. The study will also investigate the role of carnitine in insulin resistance and dyslipidemia at this same age, which may serve as grounds for future therapeutic clinical trials. Discovering genetically mediated causes of arterial stiffness or other outcomes may facilitate targeting of future therapies on susceptible youth before atherosclerotic changes are irreversible.

ELIGIBILITY:
Inclusion Criteria:

1. 11-21 year old adolescents
2. males and females
3. all ethnicities and races
4. fasting serum triglyceride levels over 130 and less than 500 mg/dL
5. fasting low density lipoprotein cholesterol (LDL-C) less than 160mg/dL.

Exclusion Criteria:

1. known seizure disorder
2. renal failure patients requiring renal replacement therapy like dialysis or renal transplant
3. diabetes mellitus type 1 or 2
4. congenital heart disease requiring surgical or catheterization intervention
5. current pregnancy or planned pregnancy during the active study participation
6. incarceration/institutionalized/wards of the state
7. known metabolic disorders that require carnitine therapy
8. nonadherence to study protocol during run-in phase defined as possessing 25% more than the expected remainder of placebo supplement pro-rated to the day of assessment

Ages: 11 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Carotid Femoral Pulse Wave Velocity | 6 months
  Carotid Femoral Pulse Wave Velocity will be measured noninvasively using applanation tonometry.

SECONDARY OUTCOMES:
Change in Fasting Triglyceride | 6 months
  Fasting serum triglycerides to be measured using conventional techniques.
Change in Insulin Resistance | 6 month
  Insulin resistance will be assessed using fasting serum glucose and fasting serum insulin to calculate homeostatic model assessment of insulin resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Justin P Zachariah, MD MPH, Principal Investigator — Study Principal Investigator
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No